CLINICAL TRIAL: NCT04776356
Title: Prospective Study to Evaluate the Continued Safety and Effectiveness of the QuickFix Small Staple to Correct Hallux Valgus Interphalangeus
Brief Title: Safety and Effectiveness of the QuickFix Small Staple
Status: Terminated | Type: Observational
Why Stopped: it was difficult to obtain subjects' consent
Sponsor: Arthrex GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AIRR-0012
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Hallux Valgus Interphalangeus
Keywords: Staple

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- QuickFix Small Staple: The QuickFix Small Staple will be used for an Akin osteotomy to correct hallux valgus interphalangeus.
  Interventions: Device: QuickFix Small Staple (Arthrex)

INTERVENTIONS:
Device: QuickFix Small Staple (Arthrex) — The Arthrex QuickFix Small Staple enables the surgeon to perform a wedge osteotomy of the first phalanx (Akin). The device is made of stainless steel and designed with barbed leg tips. The staple sizes are 8 and 10 mm wide with a 1 mm diameter.

SUMMARY:
The prospective, post-market, single-center clinical study will include 45 subjects who are candidates for surgery using the Arthrex QuickFix Small Staple for Akin osteotomy to correct hallux valgus interphalangeus. The purpose of the study is to evaluate the continued safety and effectiveness of the device. Device-related adverse events as well as patient reported outcomes (VAS, FFI, FAAM, VR-12) will be collected up to 1 year postoperative.

ELIGIBILITY:
Inclusion Criteria:

1. Subject requires surgery using the Arthrex QuickFix Small Staple for Akin osteotomy.
2. Subject is 18 years of age or older.
3. Subject is not considered a vulnerable subject (i.e. child, pregnant, nursing, prisoner, or ward of the state).
4. Subject signed informed consent and is willing and able to comply with all study requirements.

Exclusion Criteria:

1. Insufficient quantity or quality of bone.
2. Blood supply limitations and previous infections which may retard healing.
3. Foreign-body sensitivity.
4. Any active infection or blood supply limitations.
5. Conditions that tend to limit the patient's ability or willingness to restrict activities or follow directions during the healing period.
6. Subjects that are skeletally immature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 subjects, male and female, at least 18 years of age from the general population who will be treated with the Arthrex QuickFix Small Staple to correct hallux valgus interphalangeus.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Change of Visual Analogue Scale (VAS) | preoperatively, 2 weeks, 6 week, 3 months, 6 months and 12 months postoperative
  Measuring pain in the affected foot. Range 0-10 (0=best, 10=worst).
Change of Foot Function Index (FFI) | preoperatively, 3 months, 6 months and 12 months postoperative
  Measuring foot functionality. Range 0-100 (0=best, 100=worst)
Change of Foot and Ankle Ability Measure (FAAM Sport) | preoperatively, 3 months, 6 months and 12 months postoperative
  Measuring foot functionality. Range 0-100 (0=worst, 100=best)
Change of Veterans RAND 12 Iteam Health Survey (VR-12) | preoperatively, 6 months and 12 months postoperative
  Measuring quality of life. Range 0-100 (0=worst, 100=best)

CONTACTS AND LOCATIONS:
Overall Officials: Tilo Schreiter, MD, Principal Investigator — Überörtliche Gemeinschaftspraxis für Chirurgie, Unfallchirurgie, Anästhesie und Endoskopie
Locations (1):
- Überörtliche Gemeinschaftspraxis für Chirurgie, Unfallchirurgie, Anästhesie und Endoskopie, Meissen, Germany

IPD SHARING:
Plan to Share IPD: No